CLINICAL TRIAL: NCT06221345
Title: Comparison of Different Hyaluronic Acid-containing Artificial Tears on the Ocular Surface Disease in Patients With Post-cataract Surgery Dry Eye
Brief Title: Hyaluronic Acid-containing Artificial Tears in Post-cataract Surgery Dry Eye Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, CHI-CHIN-SUN, Professor, School of Medicine Chang Gung University Taoyuan, Taiwan ; Doctor, Department of Ophthalmology, Chang Gung Memorial Hospital, Keelung, Taiwan, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 60298913
Record Dates: First submitted 2024-01-02; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Dry Eye Disease; Cataract
Keywords: Hyaluronic Acid; Hydroxypropyl guar; Carboxymethylcellulose
MeSH Terms: conditions — Dry Eye Syndromes; Cataract

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HPG/HA group (Experimental): Systane HYDRATION®
  Interventions: Drug: Systane HYDRATION® Preservative-Free Lubricant Eye Drops
- CMC/HA group (Active Comparator): Optive Fusion®
  Interventions: Drug: Optive Fusion® Lubricant Eye Drops (Unit Dose)

INTERVENTIONS:
Drug: Systane HYDRATION® Preservative-Free Lubricant Eye Drops — The HPG/HA group will receive Systane HYDRATION® Preservative-Free Lubricant Eye Drops and standard of care, i.e., prednisolone acetate (Pred forte®) and levofloxacin (Cravit®), at the dosage of 1-2 drops 4 times daily for 3 weeks from Weeks 1 to 4 post-op
  Arms: HPG/HA group
Drug: Optive Fusion® Lubricant Eye Drops (Unit Dose) — The CMC/HA group will receive Optive Fusion® Lubricant Eye Drops (Unit Dose) and standard of care, i.e., prednisolone acetate (Pred forte®) and levofloxacin (Cravit®), at the dosage of 1-2 drops 4 times daily for 3 weeks from Weeks 1 to 4 post-op
  Arms: CMC/HA group

SUMMARY:
To compare the effects of hydroxypropyl guar (HPG)/hyaluronic acid (HA)- and carboxymethylcellulose (CMC)/HA-based lubricant eye drops on subjective and objective outcomes in dry eye disease (DED) patients after cataract surgery.

DETAILED DESCRIPTION:
This is a prospective, open-label, assessor-masked, interventional, randomized controlled study. A total of 70 post-cataract surgery dry-eye subjects are planned to be enrolled after eligibility confirmation at Week 1 post-operative (post-op). The subjects will then be randomized in a 1:1 ratio to either HPG/HA (Systane HYDRATION® ) or CMC/HA (Optive Fusion®) group.

From Week 1 to 3 (1st to 4th week post-op), the HPG/HA group will receive Systane HYDRATION® Preservative-Free Lubricant Eye Drops whereas the CMC/HA group will receive Optive Fusion® Lubricant Eye Drops (Unit Dose). Both groups will receive 1-2 drops of artificial tears 4 times daily for 3 weeks.

There are three visits scheduled in this study, i.e., screening, Week 1, and Week 3. The subjects will return to the study sites during these visits for efficacy and safety assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients of any race, 20 years or older who are scheduled for unilateral cataract surgery.
2. DED patients whose symptoms and signs are aggravated at baseline assessment after cataract surgery will be eligible for this study. Postoperative dry eye diagnosis criteria at baseline assessment:

   1. OSDI score >14.8* (*Eligible subject mandatory required);
   2. positive CFS* (*Eligible subject mandatory required);
   3. Schirmer's test score ≤10 mm in 5 minutes (min) (without anesthesia);
   4. TBUT ≤5 seconds (sec)

Exclusion Criteria:

1. Patients with allergy to any of the study medications, conjunctival allergy or infectious disease, history of ocular chemical or thermal burn, Stevens-Johnson syndrome or ocular pemphigoid, glaucoma or ocular hypertension, eyelid or lacrimal disease, any ocular operation within 3 months, graft-versus-host disease (GVHD), non-dry-eye ocular inflammation, trauma, or presence of uncontrolled systemic disease.
2. Before enrollment, corneal contact lens wear, history of severe systemic disease, or other conditions in the Investigator's opinion precluded enrollment.
3. Patients will be withdrawn from the study if they experience complications during surgery, or post-surgical ocular hypertension, endophthalmitis, or infectious keratitis.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-07-05 (Actual)

PRIMARY OUTCOMES:
Corneal fluorescein staining (CFS) score | Change from baseline to Weeks 1 and 3
  The CFS will be evaluated by external eye photography using the National Eye Institute (NEI) staining grid in which a score of 0 (normal) to 3 (severe) will be assigned to each of the 5 corneal regions (nasal, central, temporal, superior, and inferior). The CFS score will range between 0 and 15, and the maximum score of 15 indicates severe epitheliopathy.

SECONDARY OUTCOMES:
Ocular Surface Disease Index (OSDI) | Change from baseline to Weeks 1 and 3
  The OSDI score is a 12-item patient-reported outcomes questionnaire with an overall score ranging from 0 to 100 to assess ocular surface symptoms, and the subjects can be categorized as having a normal (0-12), mild (13-22), moderate (23-32), or severe (33-100) ocular surface disease based on their OSDI score.
Schirmer's test (without anesthesia) | Change from baseline to Weeks 1 and 3
  Schirmer's test is a quantitative test to measure maximal tear secretion capacity. A filter paper will be placed in the lower fornix for 5 min and the and the length of wetted paper is measured.While a Schirmer's test score of greater than 10 mm/5 min is classified as normal, test score of less than 5 mm/5 min indicates tear deficiency.
Tear break-up time (TBUT) | Change from baseline to Weeks 1 and 3
  TBUT is used to assess the tear film stability by recording the interval between the last blink and the first appearance of a dry spot. TBUT less than 10 sec suggests an abnormal tear film. While TBUT between 5 to 10 sec is considered marginal, TBUT less than 5 sec indicates dry eye.
Central corneal sensitivity | Change from baseline to Weeks 1 and 3
  Central corneal sensitivity will be measured using a Cochet-Bonnet esthesiometer. The 6.0-cm long nylon monofilament was held perpendicular to the subject's cornea and reduced at an interval of 0.5 cm until the subject reported that he/she was aware of the discomfort. The longer the length of the monofilament used, the greater sensitivity the subjects have.
Slit-lamp examination | Change from baseline to Weeks 1 and 3
  The slit-lamp examinations allow the physicians to identify dry eye signs on the subject. The eye structures (eyelids, cornea, and conjunctiva) of the subjects will be graded based on the United States Food and Drug Administration (FDA) grading system. While Grade 0 represents normal, the highest grade (i.e., Grade 4) indicates the subject may have very severe changes that require intervention, often medical.

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Chin Sun, M.D, Ph.D, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Keelung Chang Gung Memorial Hospital, Keelung, Taiwan

REFERENCES:
- [Derived] Sun CC, Chan YH, Huang PW, Chen NN. Evaluation of Two Artificial Tears Containing Hyaluronic Acid for Post Cataract Surgery Dry Eye Disease: A Randomized Controlled Trial. Ophthalmol Ther. 2024 Oct;13(10):2615-2627. doi: 10.1007/s40123-024-01015-9. Epub 2024 Aug 10. PMID 39127813